CLINICAL TRIAL: NCT01997099
Title: A Workflow and Satisfaction Study Evaluating the Implementation of a New "Smart" Ambulatory Infusion System: Work Smart Study
Brief Title: A Workflow and Satisfaction Study Evaluating the Implementation of a New "Smart" Ambulatory Infusion System
Acronym: Work Smart
Status: Completed | Type: Observational
Sponsor: Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Work Smart Study
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Home Healthcare Organizations Utilizing Ambulatory Infusion Pumps; Patients Requiring Infusion With an Ambulatory Infusion Pump
Keywords: Drug Library; Ambulatory Infusion Pump; Medication Safety Software; CADD®-Solis VIP; Pump Programming; Home Infusion Workflow

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Library Creation: Individuals responsible for creating the drug library
  Interventions: Device: CADD™ Solis Medication Safety Software Administrator
- Pump Programming: Individuals responsible for programming ambulatory infusion pumps
  Interventions: Device: CADD®-Solis VIP Pump
- Home Implementation: Individuals responsible for implementing ambulatory infusion pumps in patients' homes
  Interventions: Device: CADD®-Solis VIP Pump
- Workflow: Individual at the facility responsible for describing the workflow of processing and implementing an ambulatory infusion pump prior to and after introducing the CADD®-Solis VIP System.
  Interventions: Device: CADD®-Solis VIP Pump; Device: CADD™ Solis Medication Safety Software Administrator
- Ambulatory Infusion Pump Patients: Patients that receive a prescription requiring use of the CADD®-Solis VIP pump
  Interventions: Device: CADD®-Solis VIP Pump

INTERVENTIONS:
Device: CADD®-Solis VIP Pump
  Groups: Ambulatory Infusion Pump Patients; Home Implementation; Pump Programming; Workflow
Device: CADD™ Solis Medication Safety Software Administrator
  Groups: Library Creation; Workflow

SUMMARY:
The purpose of this study is to describe the home healthcare organization ambulatory infusion pump programming workflow and the process that was followed to introduce the new CADD®-Solis VIP System to each home healthcare organization or facility. In addition, this study will characterize the overall clinician (Phase 1) and patient (Phase 2) ease of use and satisfaction with the CADD®-Solis VIP System.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, post-market study conducted within the United States. There will be two independent components (Phases) to this study. Phase 1 will involve data collection to describe the home infusion pump programming workflow and the process that was used to introduce the new CADD®-Solis VIP System to each home healthcare organization. This phase is further broken down into data collection consisting of four parts: drug protocol library creation and development within the CADD™ Solis Medication Safety Software Administrator, pump programming, home care implementation, and overall workflow and new smart pump implementation. Phase 2 will involve data collection from patients that receive a prescription requiring use of the CADD®-Solis VIP pump.

ELIGIBILITY:
Phase 1

Inclusion Criteria:

* Part 1: Licensed clinicians that would be responsible for protocol library creation at the center
* Part 2: Individuals that are responsible for ambulatory infusion pump programming per the organization's standard operating procedure
* Part 3: Licensed clinicians that are responsible for performing the pump set-up and implementation activities within the home setting
* Part 4: Center personnel that are involved in the CADD®-Solis VIP System implementation process

Exclusion Criteria:

* Individuals that are unwilling or unable to answer questions as required by the protocol

Phase 2

Inclusion Criteria:

* Patients 18 years of age or older
* Patients prescribed a home infusion requiring use of the CADD®-Solis VIP pump
* Patients with infusions prescribed for a minimum duration of five (5) days
* Patient or patient's personal caregiver on behalf of the patient is willing and able to comply with the data collection requirements
* Patient is willing and able to provide informed consent for study participation

Exclusion Criteria:

* Patient is currently enrolled or plans to enroll in a concurrent study that may confound the results of this study
* Based upon a clinician's opinion, the patient has health conditions or a psychological/cognitive status that would preclude proper participation in the study and does not have a personal caregiver available to perform study activities on behalf of the patient
* Previous use or experience with the CADD®-Solis VIP pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Home healthcare organizations that utilize ambulatory infusion pumps for their patients will be approached for participation in the study
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Protocol Library Creation | 2-6 weeks post-enrollment
  Characterize the effort required to create a new drug protocol library
Describe Library Protocols and Safety Limits Utilized | 2-6 weeks post-enrollment
  Summarize the drug protocols that were created in the library and describe the soft and hard safety limits that were utilized
Pump Programming Ease of Use | Day 1 - Immediately post-enrollment
  Characterize the ease of use associated with programming the CADD®-Solis VIP pump
Pump Programming Errors | Day 1 - Immediately post-enrollment
  Summarize and describe any possible programming errors
Patient Training and Pump Set-up | 2-4 months post-enrollment
  Characterize the home health nurse perception of patient training and pump set-up within the home
Characterize Training Time for the New Pump System | 2-4 months post-enrollment
  Describe the training time associated with implementing a new ambulatory infusion pump in each step of a home healthcare organization's workflow
Workflow Changes | 2-4 months post-enrollment
  Characterize the workflow changes that need to be implemented at home healthcare organizations when adopting the CADD®-Solis VIP System
Overall Patient/Caregiver Satisfaction with the Pump | 5-7 Days Post-Enrollment
  Assess the overall patient/personal caregiver satisfaction with the CADD®-Solis VIP pump

SECONDARY OUTCOMES:
Number of Alarms Reported | 5-7 Days Post-Enrollment
  Summarize the number of alarms reported
Alarm Troubleshooting | 5-7 Days Post-Enrollment
  Quantify the ability of the patient or caregiver to successfully troubleshoot the alarms
Pump Difficulties | 5-7 Days Post-Enrollment
  Characterize any difficulties experienced with use of the pump
Pump Ease of Use | 5-7 Days Post-Enrollment
  Characterize the ease of use of the pump

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Brown, MBA, PharmD, Principal Investigator — Thomas Jefferson University Hospital - Jefferson Home Infusion
Locations (2):
- United States (2):
  - Big Sky IV Care, Kalispell, Montana
  - Thomas Jefferson University Hospital - Jefferson Home Infusion, Philadelphia, Pennsylvania